CLINICAL TRIAL: NCT07243613
Title: Acute Psychoneuroendocrine Responses to Maximal Exertion Following High-Load Training in Elite Rowers: A Sex-Based Comparative Study
Brief Title: Pre-Exercise Mood and Physiological Responses to Maximal Effort in Elite Rowers
Acronym: 6000MFPOMS2024
Status: Completed | Type: Observational
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Other Study IDs: RowersPOMS20236000
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2024-03

CONDITIONS: Health Adult Subjects
Keywords: Exercise-induced Fatigue; Elithe Athletes; Neurtransmitters; Mood State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elite male rowers
  Interventions: Other: Maximal Rowing Test
- Elite female rowers
  Interventions: Other: Maximal Rowing Test

INTERVENTIONS:
Other: Maximal Rowing Test — Participants completed a 2000-meter maximal rowing ergometer test on day 8 following a standardized 7-day high-load training period. The test served as the physiological and psychological stressor used to assess acute fatigue responses.

SUMMARY:
This study examined how the body and mood respond to intense physical effort in elite male and female rowers. Athletes completed a maximal rowing test after one week of hard training. Researchers collected blood samples before and after exercise to measure stress hormones and brain-related chemicals. They also used a short questionnaire to assess how the athletes felt emotionally before the test. The goal of the study is to better understand how physical and mental fatigue develop in well-trained athletes, and whether men and women respond differently.

DETAILED DESCRIPTION:
This observational cohort study was designed to characterize acute physiological and psychological responses to maximal exertion following a high-load training period in elite male and female rowers. The main aim was to investigate how accumulated training fatigue affects hormonal and neurochemical responses to intense effort, and whether these responses differ by sex.

Participants were national-level athletes undergoing a standardized 7-day training camp, during which they completed identical high-intensity training sessions. On day 8, all participants performed a 2000-m maximal rowing ergometer test under controlled conditions. Blood samples were collected at three time points: before exercise (PRE), immediately post-exercise (POST), and 1 hour post-exercise (1H).

Biomarkers analyzed in serum included cortisol, total testosterone, serotonin (5-HT), dopamine (DA), gamma-aminobutyric acid (GABA), and tryptophan. The testosterone-to-cortisol (T/C) ratio was used as an index of anabolic-catabolic balance, while the 5-HT/DA ratio was examined as a neurochemical indicator of central fatigue.

In parallel, mood state was assessed once prior to the exertion test using the standardized Profile of Mood States (POMS) questionnaire. This provided insight into psychological readiness and emotional state entering maximal effort.

A total of 28 athletes (12 females, 16 males) completed the full protocol. There were no missing data. The study did not involve any interventions, randomization, or masking. Statistical analyses included repeated-measures ANOVA for time and group effects, and calculation of within-group effect sizes (Cohen's d).

Although no biospecimens were retained beyond initial analysis, serum samples were processed and stored short-term according to laboratory standards. The study followed ethical approval procedures and informed consent was obtained from all participants. No external monitoring, third-party auditing, or source data verification was implemented, as this was a single-site, non-interventional academic study.

The data collected provide a multidimensional profile of physiological and mood-related responses to intense physical effort under conditions of cumulative fatigue. These findings may inform future monitoring strategies in high-performance sport and support individualized recovery planning.

ELIGIBILITY:
Inclusion Criteria:

Aged 19-25 years National-level competitive rower Minimum 5 years of structured rowing training Currently in full training and competition season Completed 7-day standardized high-load training program Provided written informed consent

Exclusion Criteria:

Use of medications or supplements affecting hormonal or neurochemical markers Known endocrine, neurological, or psychiatric disorders Injury or illness interfering with training or testing Incomplete participation in the training camp or testing protocol

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All participants were recruited and tested at the Central Sports Centre - Olympic Preparation Center (COS OPO) in Wałcz, Poland, during a national team training camp under standardized conditions.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Serum Testosterone concentration | Before exercise, immediately after, and 1 hour after recovery
  Testosterone concentration will be measured in serum using immunoassay. Units: ng/mL.
Serum Cortisol concentration | Before exercise, immediately after, and 1 hour after recovery
  Cortisol concentration will be measured in serum using an immunoassay. Units: ng/mL
Serum Serotonin concentration | Before exercise, immediately after, and 1 hour after recovery
  Serotonin concentration will be measured in serum using an immunoassay. Units: ng/mL
Serum Gamma-aminobutyric acid (GABA) concentration | Before exercise, immediately after, and 1 hour after recovery
  GABA concentration will be measured in serum using an immunoassay. Units: µg/dL
Serum Tryptophan concentration | Before exercise, immediately after, and 1 hour after recovery
  Tryptophan concentration will be measured in serum using an immunoassay. Units: µg/dL
Profile of Mood States | Before exercise
  Self-reported mood assessed using the Profile of Mood States (POMS); total and subscale scores.

SECONDARY OUTCOMES:
T:C ratio | Before exercise, immediately after, and 1 hour after recovery
  Ratio of serum testosterone to cortisol as an index of anabolic-catabolic balance
S:D ratio | Before exercise, immediately after, and 1 hour after recovery
  Ratio of serum serotonin to dopamine to assess neurochemical fatigue profile.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Skarpańska-Stejborn, Professor, Study Director — Poznań University of Physical Education, Faculty of Sport Sciences in Gorzów Wielkopolski, Poland;
Locations (1):
- Poznań University of Physical Education, Poznan, Greater Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Data will be used only for internal analysis and dissemination in scientific publications in aggregate form, in accordance with ethical approval.